

## **STUDY SYNOPSIS**

| Study title | MULTICENTER, NON-INTERVENTIONAL STUDY, DESCRIBING PATIENTS WITH INHERITED RETINAL DISEASE (IRD) IN FRANCE |
|---|---|
| Short title | EPI-GenRet |
| Sponsor | Strasbourg University Hospitals |
| Coordinating/Principal Investigator | Pr Hélène DOLLFUS |
| Collaborative partner | Novartis Pharma SAS |
| HUS n° | 8173 |
| ID RCB n° | 2021-A01786-35 |
| NCT | NCT05122442 |
| Study rationale | Genetic diagnostic testing becomes increasingly important for enhancing our understanding of the disease notably the genetics and providing the best care to the patients ("Recommendations on Clinical Assessment of Patients with Inherited Retinal Degenerations - 2016," 2016), and several initiatives seek to gather more data in order to better understand and treat those diseases. Within this context, Novartis and SENSGENE/Strasbourg University Hospitals (HUS) want to set up, through a research collaboration, a non-interventional study in France to better understand the epidemiology of IRDs, particularly the distribution of pathogenic variants in patients. This study aims to serve as a starter study to implement an IRD national registry led by SENSGENE/Strasbourg University Hospitals (HUS). The data collected might also be used to populate global European registries (cf ERN-EYE initiatives). The primary objective has been defined in a sufficient broad way to address this perspective of registries. As IRDs can present from birth to late middle age, this study will include both children and adult patients regardless of age, sex, and the type of IRD. |
| | The primary objective of this study is to describe the type of IRD of |
| Primary Objective | patients clinically diagnosed and who attended a consultation at |
| Trimary Objective | one of participating centers from SENSGENE network over the |
| Secondary Objectives | inclusion period. The secondary objectives are stated for patients with IRD who attended a consultation at one of the participating centers from SENSGENE network over the inclusion period. • To describe the genetic diagnosis • To describe the genetic testing characteristics • To describe the distribution of genes and pathogenic variants (class 4 and class 5) associated with IRDs • To describe the distribution of variant of uncertain significance (VUS - class 3 variants) in IRD-associated genes • To describe the proportion of unsolved patients • To describe the type of pathogenic variants in each IRD-associated gene identified |



| Proportion of patients by type of analysis performed for definitive molecular genetic diagnosis Proportion of each type of genetic analysis performed and duration between clinical diagnosis and definitive molecular genetic diagnosis Proportion of genes with at least 1 pathogenic variant identified (classified as class 4 likely pathogenic and class 5 pathogenic) according to transmission mode Proportion of variants according to their classification (class 4 and 5) in a specific gene and in all IRD genes Proportion of variants of uncertain significance (VUS-class 3 variants) Proportion of unsolved patients Proportion of pathogenic variants according to the: Mutation's nomenclature Nature of gene mutation Allelic status | | To evaluate the potential correlation between the patient's |
|---|---|---|
| To describe the diagnosis pathway To describe the socio-demographic characteristics of patients To describe the socio-demographic characteristics of patients To describe the therapeutic care of patients Proportion of patients by type of IRD (based on ORPHA classification for IRD) Proportion of patients by type of analysis performed for definitive molecular genetic diagnosis Proportion of each type of genetic analysis performed and duration between clinical diagnosis and definitive molecular genetic diagnosis Proportion of genes with at least 1 pathogenic variant identified (classified as class 4 likely pathogenic and class 5 pathogenic) according to transmission mode Proportion of variants according to their classification (class 4 and 5) in a specific gene and in all IRD genes Proportion of variants of uncertain significance (VUS-class 3 variants) Proportion of variants of uncertain significance (VUS-class 3 variants) Proportion of pathogenic variants according to the: Mutation's nomenclature Nature of gene mutation Allelic status Origin of the allele Proportion of patient with family segregation assessment Proportion of similar genotype in other family members Proportion of "classic cases", i.e. patients whose clinical phenotype is associated with the expected genotype Proportion of patients whose type of IRD (ORPHA classification) was modified after definitive molecular genetic diagnosis Proportion of patients by: Age at first symptom onset Circumstances of discovery Type of clinical assessments to confirm the clinical diagnosis Age at date of clinical diagnosis | | |
| Primary endpoint • To describe the socio-demographic characteristics of patients • To describe the therapeutic care of patients Proportion of patients by type of IRD (based on ORPHA classification for IRD) • Proportion of patients by type of analysis performed for definitive molecular genetic diagnosis • Proportion of each type of genetic analysis performed and duration between clinical diagnosis and definitive molecular genetic diagnosis • Proportion of genes with at least 1 pathogenic variant identified (classified as class 4 likely pathogenic and class 5 pathogenic) according to transmission mode • Proportion of variants according to their classification (class 4 and 5) in a specific gene and in all IRD genes • Proportion of variants of uncertain significance (VUS-class 3 variants) • Proportion of variants of uncertain significance (VUS-class 3 variants) • Proportion of pathogenic variants according to the: • Mutation's nomenclature • Nature of gene mutation • Allelic status • Origin of the allele • Proportion of patient with family segregation assessment • Proportion of similar genotype in other family members • Proportion of "classic cases", i.e. patients whose clinical phenotype is associated with unusual/unexpected genotype • Proportion of "atypic cases", i.e. patients whose clinical phenotype is associated with unusual/unexpected genotype • Proportion of patients whose type of IRD (ORPHA classification) was modified after definitive molecular genetic diagnosis • Proportion of patients by: • Age at first symptom onset • Circumstances of discovery • Type of clinical assessments to confirm the clinical diagnosis • Age at date of clinical diagnosis | | To describe the clinical characteristics |
| patients To describe the therapeutic care of patients Proportion of patients by type of IRD (based on ORPHA classification for IRD) Proportion of patients by type of analysis performed for definitive molecular genetic diagnosis Proportion of each type of genetic analysis performed and duration between clinical diagnosis and definitive molecular genetic diagnosis Proportion of genes with at least 1 pathogenic variant identified (classified as class 4 likely pathogenic and class 5 pathogenic) according to transmission mode Proportion of variants according to their classification (class 4 and 5) in a specific gene and in all IRD genes Proportion of variants of uncertain significance (VUS-class 3 variants) Proportion of unsolved patients Proportion of unsolved patients Proportion of pathogenic variants according to the: Mutation's nomenclature Nature of gene mutation Allelic status Origin of the allele Proportion of similar genotype in other family members Proportion of "classic cases", i.e. patients whose clinical phenotype is associated with the expected genotype Proportion of "atypic cases", i.e. patients whose clinical phenotype is associated with the expected genotype Proportion of matients whose type of IRD (ORPHA classification) was modified after definitive molecular genetic diagnosis Proportion of patients by: Age at first symptom onset Circumstances of discovery Type of clinical assessments to confirm the clinical diagnosis Age at date of clinical diagnosis | | <ul> <li>To describe the diagnosis pathway</li> </ul> |
| Primary endpoint Proportion of patients by type of IRD (based on ORPHA classification for IRD) • Proportion of patients by type of analysis performed for definitive molecular genetic diagnosis • Proportion of each type of genetic analysis performed and duration between clinical diagnosis and definitive molecular genetic diagnosis • Proportion of genes with at least 1 pathogenic variant identified (classified as class 4 likely pathogenic and class 5 pathogenic) according to transmission mode • Proportion of variants according to their classification (class 4 and 5) in a specific gene and in all IRD genes • Proportion of variants of uncertain significance (VUS-class 3 variants) • Proportion of variants of uncertain significance (VUS-class 3 variants) • Proportion of pathogenic variants according to the: • Mutation's nomenclature • Nature of gene mutation • Allelic status • Origin of the allele • Proportion of patient with family segregation assessment • Proportion of similar genotype in other family members • Proportion of similar genotype in other family members • Proportion of "classic cases", i.e. patients whose clinical phenotype is associated with the expected genotype • Proportion of "atypic cases", i.e. patients whose clinical phenotype is associated with unusual/unexpected genotype • Proportion of patients whose type of IRD (ORPHA classification) was modified after definitive molecular genetic diagnosis • Proportion of patients by: • Age at first symptom onset • Circumstances of discovery • Type of clinical assessments to confirm the clinical diagnosis • Age at date of clinical diagnosis | | |
| Proportion of patients by type of IRD (based on ORPHA classification for IRD) Proportion of patients by type of analysis performed for definitive molecular genetic diagnosis Proportion of each type of genetic analysis performed and duration between clinical diagnosis and definitive molecular genetic diagnosis Proportion of genes with at least 1 pathogenic variant identified (classified as class 4 likely pathogenic and class 5 pathogenic) according to transmission mode Proportion of variants according to their classification (class 4 and 5) in a specific gene and in all IRD genes Proportion of variants of uncertain significance (VUS-class 3 variants) Proportion of variants of uncertain significance (VUS-class 3 variants) Proportion of pathogenic variants according to the: Mutation's nomenclature Nature of gene mutation Allelic status Origin of the allele Proportion of patient with family segregation assessment Proportion of similar genotype in other family members Proportion of "classic cases", i.e. patients whose clinical phenotype is associated with the expected genotype Proportion of "atypic cases", i.e. patients whose clinical phenotype is associated with unusual/unexpected genotype Proportion of patients whose type of IRD (ORPHA classification) was modified after definitive molecular genetic diagnosis Proportion of patients by: Age at first symptom onset Circumstances of discovery Type of clinical assessments to confirm the clinical diagnosis Age at date of clinical diagnosis | | · · |
| Frimary enapoint Proportion of patients by type of analysis performed for definitive molecular genetic diagnosis Proportion of each type of genetic analysis performed and duration between clinical diagnosis and definitive molecular genetic diagnosis Proportion of genes with at least 1 pathogenic variant identified (classified as class 4 likely pathogenic and class 5 pathogenic) according to transmission mode Proportion of variants according to their classification (class 4 and 5) in a specific gene and in all IRD genes Proportion of variants of uncertain significance (VUS-class 3 variants) Proportion of unsolved patients Proportion of pathogenic variants according to the: Mutation's nomenclature Nature of gene mutation Allelic status Origin of the allele Proportion of patient with family segregation assessment Proportion of similar genotype in other family members Proportion of "classic cases", i.e. patients whose clinical phenotype is associated with unusual/unexpected genotype Proportion of "atypic cases", i.e. patients whose clinical phenotype is associated with unusual/unexpected genotype Proportion of patients whose type of IRD (ORPHA classification) was modified after definitive molecular genetic diagnosis Proportion of patients by: Age at first symptom onset Circumstances of discovery Type of clinical assessments to confirm the clinical diagnosis Age at date of clinical diagnosis | | |
| definitive molecular genetic diagnosis Proportion of each type of genetic analysis performed and duration between clinical diagnosis and definitive molecular genetic diagnosis Proportion of genes with at least 1 pathogenic variant identified (classified as class 4 likely pathogenic and class 5 pathogenic) according to transmission mode Proportion of variants according to their classification (class 4 and 5) in a specific gene and in all IRD genes Proportion of variants of uncertain significance (VUS-class 3 variants) Proportion of unsolved patients Proportion of pathogenic variants according to the: Mutation's nomenclature Nature of gene mutation Allelic status Origin of the allele Proportion of patient with family segregation assessment Proportion of similar genotype in other family members Proportion of "classic cases", i.e. patients whose clinical phenotype is associated with the expected genotype Proportion of "atypic cases", i.e. patients whose clinical phenotype is associated with unusual/unexpected genotype Proportion of patients whose type of IRD (ORPHA classification) was modified after definitive molecular genetic diagnosis Proportion of patients by: Age at first symptom onset Circumstances of discovery Type of clinical diagnosis Age at date of clinical diagnosis | Primary endpoint | |
| duration between clinical diagnosis and definitive molecular genetic diagnosis Proportion of genes with at least 1 pathogenic variant identified (classified as class 4 likely pathogenic and class 5 pathogenic) according to transmission mode Proportion of variants according to their classification (class 4 and 5) in a specific gene and in all IRD genes Proportion of variants of uncertain significance (VUS-class 3 variants) Proportion of unsolved patients Proportion of pathogenic variants according to the: Mutation's nomenclature Nature of gene mutation Allelic status Origin of the allele Proportion of patient with family segregation assessment Proportion of similar genotype in other family members Proportion of "classic cases", i.e. patients whose clinical phenotype is associated with the expected genotype Proportion of "atypic cases", i.e. patients whose clinical phenotype is associated with unusual/unexpected genotype Proportion of patients whose type of IRD (ORPHA classification) was modified after definitive molecular genetic diagnosis Proportion of patients by: Age at first symptom onset Circumstances of discovery Type of clinical diagnosis Age at date of clinical diagnosis | | |
| (classified as class 4 likely pathogenic and class 5 pathogenic) according to transmission mode Proportion of variants according to their classification (class 4 and 5) in a specific gene and in all IRD genes Proportion of variants of uncertain significance (VUS-class 3 variants) Proportion of unsolved patients Proportion of pathogenic variants according to the: Mutation's nomenclature Nature of gene mutation Allelic status Origin of the allele Proportion of patient with family segregation assessment Proportion of similar genotype in other family members Proportion of "classic cases", i.e. patients whose clinical phenotype is associated with the expected genotype Proportion of "atypic cases", i.e. patients whose clinical phenotype is associated with unusual/unexpected genotype Proportion of patients whose type of IRD (ORPHA classification) was modified after definitive molecular genetic diagnosis Proportion of patients by: Age at first symptom onset Circumstances of discovery Type of clinical assessments to confirm the clinical diagnosis Age at date of clinical diagnosis | | duration between clinical diagnosis and definitive molecular |
| and 5) in a specific gene and in all IRD genes Proportion of variants of uncertain significance (VUS-class 3 variants) Proportion of unsolved patients Proportion of pathogenic variants according to the: Mutation's nomenclature Nature of gene mutation Allelic status Origin of the allele Proportion of patient with family segregation assessment Proportion of similar genotype in other family members Proportion of "classic cases", i.e. patients whose clinical phenotype is associated with the expected genotype Proportion of "atypic cases", i.e. patients whose clinical phenotype is associated with unusual/unexpected genotype Proportion of patients whose type of IRD (ORPHA classification) was modified after definitive molecular genetic diagnosis Proportion of patients by: Age at first symptom onset Circumstances of discovery Type of clinical assessments to confirm the clinical diagnosis Age at date of clinical diagnosis | | (classified as class 4 likely pathogenic and class 5 pathogenic) |
| variants) Proportion of unsolved patients Proportion of pathogenic variants according to the: Mutation's nomenclature Nature of gene mutation Allelic status Origin of the allele Proportion of patient with family segregation assessment Proportion of similar genotype in other family members Proportion of "classic cases", i.e. patients whose clinical phenotype is associated with the expected genotype Proportion of "atypic cases", i.e. patients whose clinical phenotype is associated with unusual/unexpected genotype Proportion of patients whose type of IRD (ORPHA classification) was modified after definitive molecular genetic diagnosis Proportion of patients by: Age at first symptom onset Circumstances of discovery Type of clinical assessments to confirm the clinical diagnosis Age at date of clinical diagnosis | | |
| Proportion of pathogenic variants according to the: Mutation's nomenclature Nature of gene mutation Allelic status Origin of the allele Proportion of patient with family segregation assessment Proportion of similar genotype in other family members Proportion of "classic cases", i.e. patients whose clinical phenotype is associated with the expected genotype Proportion of "atypic cases", i.e. patients whose clinical phenotype is associated with unusual/unexpected genotype Proportion of patients whose type of IRD (ORPHA classification) was modified after definitive molecular genetic diagnosis Proportion of patients by: Age at first symptom onset Circumstances of discovery Type of clinical assessments to confirm the clinical diagnosis Age at date of clinical diagnosis | | |
| O Mutation's nomenclature Nature of gene mutation Allelic status Origin of the allele Proportion of patient with family segregation assessment Proportion of similar genotype in other family members Proportion of "classic cases", i.e. patients whose clinical phenotype is associated with the expected genotype Proportion of "atypic cases", i.e. patients whose clinical phenotype is associated with unusual/unexpected genotype Proportion of patients whose type of IRD (ORPHA classification) was modified after definitive molecular genetic diagnosis Proportion of patients by: Age at first symptom onset Circumstances of discovery Type of clinical assessments to confirm the clinical diagnosis Age at date of clinical diagnosis | | Proportion of unsolved patients |
| O Nature of gene mutation Allelic status Origin of the allele Proportion of patient with family segregation assessment Proportion of similar genotype in other family members Proportion of "classic cases", i.e. patients whose clinical phenotype is associated with the expected genotype Proportion of "atypic cases", i.e. patients whose clinical phenotype is associated with unusual/unexpected genotype Proportion of patients whose type of IRD (ORPHA classification) was modified after definitive molecular genetic diagnosis Proportion of patients by: Age at first symptom onset Circumstances of discovery Type of clinical assessments to confirm the clinical diagnosis Age at date of clinical diagnosis | | Proportion of pathogenic variants according to the: |
| <ul> <li>Proportion of patient with family segregation assessment</li> <li>Proportion of similar genotype in other family members</li> <li>Proportion of "classic cases", i.e. patients whose clinical phenotype is associated with the expected genotype</li> <li>Proportion of "atypic cases", i.e. patients whose clinical phenotype is associated with unusual/unexpected genotype</li> <li>Proportion of patients whose type of IRD (ORPHA classification) was modified after definitive molecular genetic diagnosis</li> <li>Proportion of patients by: <ul> <li>Age at first symptom onset</li> <li>Circumstances of discovery</li> <li>Type of clinical assessments to confirm the clinical diagnosis</li> <li>Age at date of clinical diagnosis</li> </ul> </li> </ul> | Secondary endpoints | <ul><li>Nature of gene mutation</li><li>Allelic status</li></ul> |
| <ul> <li>Proportion of "classic cases", i.e. patients whose clinical phenotype is associated with the expected genotype</li> <li>Proportion of "atypic cases", i.e. patients whose clinical phenotype is associated with unusual/unexpected genotype</li> <li>Proportion of patients whose type of IRD (ORPHA classification) was modified after definitive molecular genetic diagnosis</li> <li>Proportion of patients by: <ul> <li>Age at first symptom onset</li> <li>Circumstances of discovery</li> <li>Type of clinical assessments to confirm the clinical diagnosis</li> <li>Age at date of clinical diagnosis</li> </ul> </li> </ul> | | |
| <ul> <li>phenotype is associated with the expected genotype</li> <li>Proportion of "atypic cases", i.e. patients whose clinical phenotype is associated with unusual/unexpected genotype</li> <li>Proportion of patients whose type of IRD (ORPHA classification) was modified after definitive molecular genetic diagnosis</li> <li>Proportion of patients by: <ul> <li>Age at first symptom onset</li> <li>Circumstances of discovery</li> <li>Type of clinical assessments to confirm the clinical diagnosis</li> <li>Age at date of clinical diagnosis</li> </ul> </li> </ul> | | Proportion of similar genotype in other family members |
| <ul> <li>phenotype is associated with unusual/unexpected genotype</li> <li>Proportion of patients whose type of IRD (ORPHA classification) was modified after definitive molecular genetic diagnosis</li> <li>Proportion of patients by: <ul> <li>Age at first symptom onset</li> <li>Circumstances of discovery</li> <li>Type of clinical assessments to confirm the clinical diagnosis</li> <li>Age at date of clinical diagnosis</li> </ul> </li> </ul> | | |
| <ul> <li>was modified after definitive molecular genetic diagnosis</li> <li>Proportion of patients by: <ul> <li>Age at first symptom onset</li> <li>Circumstances of discovery</li> <li>Type of clinical assessments to confirm the clinical diagnosis</li> <li>Age at date of clinical diagnosis</li> </ul> </li> </ul> | | |
| <ul> <li>Age at first symptom onset</li> <li>Circumstances of discovery</li> <li>Type of clinical assessments to confirm the clinical diagnosis</li> <li>Age at date of clinical diagnosis</li> </ul> | | |
| <ul> <li>Circumstances of discovery</li> <li>Type of clinical assessments to confirm the clinical diagnosis</li> <li>Age at date of clinical diagnosis</li> </ul> | | Proportion of patients by: |
| <ul> <li>Circumstances of discovery</li> <li>Type of clinical assessments to confirm the clinical diagnosis</li> <li>Age at date of clinical diagnosis</li> </ul> | | <ul> <li>Age at first symptom onset</li> </ul> |
| <ul> <li>Type of clinical assessments to confirm the clinical diagnosis</li> <li>Age at date of clinical diagnosis</li> </ul> | | |
| <ul> <li>Age at date of clinical diagnosis</li> </ul> | | o Type of clinical assessments to confirm the clinical |
| | | _ |
| <ul> <li>Type and number of current symptoms related to</li> </ul> | | |
| IRD at consultation | | |
| <ul> <li>Associated clinical signs</li> </ul> | | <ul> <li>Associated clinical signs</li> </ul> |



| | <ul> <li>Medical history of interest</li> <li>Proportion of patients according to the values of visual acuity</li> </ul> |
|---|---|
| | (VA) and visual field (VF) by patients' clinical characteristics |
| | Proportion of patients with a cystoid macular oedema (CME) on<br>last coherence tomography (OCT) done |
| | Proportion of patients with preserved macular area appearance<br>by autofluorescence at consultation |
| | Proportion of patients according to lens status |
| | Proportion of patients with cataract at consultation |
| | Proportion of patients with posterior capsular opacification |
| | Proportion of patients with cataract (phakic and pseudophakic) with an impact on VA |
| | Proportion of patients by type of clinical assessments performed |
| | Diagnostic odyssey (Length of time from the first symptoms onset to the clinical diagnosis and Length of time from the previous molecular genetic test and the definitive molecular genetic diagnosis for patient who already had a molecular genetic test) |
| | Proportion of patients by age class, gender, type of occupation and geographical origin |
| | Proportion of patients by type of treatments administered for IRD |
| | This study is a multicenter, cross-sectional non-interventional study that aims to set up a registry of patients with IRD in France. |
| Study design | This study relies on primary data collection and a cross sectional design. Data will be collected for both patients with prevalent IRD (patients who were already clinically diagnosed with IRD before the inclusion in the study) and patients with incident IRD (patients who were clinically diagnosed with IRD upon their inclusion in the study). To address the primary objective, all patients seen by the physician over the inclusion period following site initiation will be included into the study, on a consecutive and exhaustive basis until a maximum of 1000 patients is reached (registry starter). |
| . 5 | Given the capacity of sites to screen patients over one year (around 3000 patients), the inclusion of patients into the study will be limited to the first 1000 patients in order to favor the data collection quality by limiting the sites workload. This will also encourage the inclusion of the patients exhaustively, especially for high volume sites for which this registry represents a deep work. However, it should be reminded that this study is a starter study that is planned to be extended to a larger national registry. |
| | Since this study is non-interventional, nor clinical interventions neither genetic tests, imaging and assessment schedule will be |



| physicians' routine practice. Patients included in this study must have either available geneti results upon their inclusion in the study (whether the result of thi test is positive or negative) or a genetic testing prescription for IRI (genetic testing through PFMG platform or from a traditions reference public laboratory). Given the delay for obtaining geneti results, the data may be available within approximately 12 month after the test prescription. Only the patients who meet all the following inclusion criteria can be included in this study: • All patients, whatever age or gender, clinically diagnose with IRD or with high suspicion for IRDs based on clinical examination and functional tests (such as fundus exam an ERG), regardless of genetic testing • Patients who attended a consultation at one of the participating centers from SENSGENE network over the inclusion period starting from sites initiation • Patients who attended a consultation at one of the participating centers from SENSGENE network over the inclusion period starting from sites initiation • Patients who had been prescribed a genetic test for IRD priot to or at the date of inclusion. • Patients who had been prescribed a genetic test for IRD priot to or at the date of inclusion. • Patients/Parents/Legally authorized representatives (LAR opposed to the collection and processing of their medical data of their children/the | | required as part of this study, and all data will be collected as per |
|---|---|---|
| Patients included in this study must have either available genetic results upon their inclusion in the study (whether the result of this test is positive or negative) or a genetic testing prescription for IRI (genetic testing through PFMG platform or from a traditional reference public laboratory). Given the delay for obtaining genetic results, the data may be available within approximately 12 month after the test prescription. Only the patients who meet all the following inclusion criteria can be included in this study: • All patients, whatever age or gender, clinically diagnose with IRD or with high suspicion for IRDs based on clinics examination and functional tests (such as fundus exam an ERG), regardless of genetic testing • Patients who attended a consultation at one of the participating centers from SENSGENE network over the inclusion period starting from sites initiation • Patients who attended a consultation at one of the participating centers from SENSGENE network over the inclusion period starting from sites initiation • Patients who attended a consultation at one of the participating centers from SENSGENE network over the inclusion period starting from sites initiation • Patients who are suffering from sites initiation • Patients who present at least one of the following non-inclusion criteria cannot be included in this study: • Patients/Parents/Legally authorized representatives (LAR opposed to the collection and processing of their medica data/the medical data of their children/the medical data of the person for whom they are LAR; • Patients who are suffering from any other retinal disorder on optic neuropathy that may clinically or genetically overlay with IRD or non-genetic (phenocopy); • Patients/parents/Legally authorized representatives (LAR refusing genetic testing; • Patients/parents/Legally authorized representatives (LAR refusing genetic testing; • Patients/parents/Legally authorized representatives (LAR refusing genetic testing; • Patients who are suffering from any other re | | |
| (genetic testing through PFMG platform or from a traditional reference public laboratory). Given the delay for obtaining genetic results, the data may be available within approximately 12 month after the test prescription. Only the patients who meet all the following inclusion criteria can be included in this study: | | Patients included in this study must have either available genetic results upon their inclusion in the study (whether the result of this test is positive or negative) or a genetic testing prescription for IRE |
| reference public laboratory). Given the delay for obtaining genetic results, the data may be available within approximately 12 month after the test prescription. Only the patients who meet all the following inclusion criteria can be included in this study: • All patients, whatever age or gender, clinically diagnose with IRD or with high suspicion for IRDs based on clinical examination and functional tests (such as fundus exam an ERG), regardless of genetic testing • Patients who attended a consultation at one of the participating centers from SENSGENE network over the inclusion period starting from sites initiation • Patients who had been prescribed a genetic test for IRD prior to or at the date of inclusion. • Patients who had been prescribed a genetic test for IRD prior to or at the date of inclusion. • Patients who present at least one of the following non-inclusion criteria cannot be included in this study: • Patients/Parents/Legally authorized representatives (LAR opposed to the collection and processing of their medical data/the medical data of their children/the medical data/the medical data of their children/the medical data/the medical data of their children/the medical data of the person for whom they are LAR; • Patients who are suffering from any other retinal disorder of optic neuropathy that may clinically or genetically overlay with IRD or non-genetic (phenocopy); • Patients have a suffering from any other retinal disorder of optic neuropathy that may clinically or genetically overlay with IRD or non-genetic (phenocopy); • Patients lacking decision-making capacity: Menta incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation. French reference and competence centers for rare eye diseases and gathered within the SENSGENE network. The Filière de sant maladies rares (FSMR) SENSGENE futfills national missions around rare sensory diseases with the aim of improving the care of patients coordinating and encouraging research and developing training and i | | |
| results, the data may be available within approximately 12 month after the test prescription. Only the patients who meet all the following inclusion criteria can be included in this study: • All patients, whatever age or gender, clinically diagnose with IRD or with high suspicion for IRDs based on clinical examination and functional tests (such as fundus exam an ERG), regardless of genetic testing • Patients who attended a consultation at one of the participating centers from SENSGENE network over the inclusion period starting from sites initiation • Patients who had been prescribed a genetic test for IRD priod to or at the date of inclusion. Patients who present at least one of the following non-inclusion criteria cannot be included in this study: • Patients/Parents/Legally authorized representatives (LAR opposed to the collection and processing of their medical data/the medical data of their children/the medical data of their children/the medical data of their children/the medical data of the person for whom they are LAR; • Patients who are suffering from any other retinal disorder on optic neuropathy that may clinically or genetically overlay with IRD or non-genetic (phenocopy); • Patients/parents/Legally authorized representatives (LAR refusing genetic testing; • Patients lacking decision-making capacity; Menta incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation. French reference and competence centers for rare eye diseases and gathered within the SENSGENE fulfills national missions around rare sensory diseases with the aim of improving the care of patients coordinating and encouraging research and developing training and information. Seven French reference and competence centers for rare eye diseases: HU-Necker-Enfants Malades-APPH (Paris), CHNO XV-XX (Paris), CHI Créteil, HU Strasbourg, CHU Montpeller. • Two competence centers for rare eye diseases: CHU Nantes and CHU Lille This study will set up a registry that will include all eligible patient wit | | reference public laboratory). Given the delay for obtaining gener |
| Only the patients who meet all the following inclusion criteria can be included in this study: • All patients, whatever age or gender, clinically diagnose with IRD or with high suspicion for IRDs based on clinica examination and functional tests (such as fundus exam an ERG), regardless of genetic testing • Patients who attended a consultation at one of the participating centers from SENSGENE network over the inclusion period starting from Sites initiation • Patients who had been prescribed a genetic test for IRD prior to or at the date of inclusion. • Patients who present at least one of the following non-inclusion criteria cannot be included in this study: • Patients/Parents/Legally authorized representatives (LAR opposed to the collection and processing of their medical data of their children/the medical data of their children/the medical data of their children/the medical data of the person for whom they are LAR; • Patients who are suffering from any other retinal disorder on optic neuropathy that may clinically or genetically overlal with IRD or non-genetic (phenocopy); • Patients/parents/Legally authorized representatives (LAR refusing genetic testing; • Patients lacking decision-making capacity: Menta incapacity, unwillingness, or language barriers precludin adequate understanding or cooperation. French reference and competence centers for rare eye diseases an gathered within the SENSGENE network. The Filière de sant maladies rares (FSMR) SENSGENE network will be contacted to participate in the study. Conduct of the study • Five c | | |
| included in this study: All patients, whatever age or gender, clinically diagnose with IRD or with high suspicion for IRDs based on clinical examination and functional tests (such as fundus exam an ERG), regardless of genetic testing Patients who attended a consultation at one of the participating centers from SENSGENE network over the inclusion period starting from sites initiation Patients who had been prescribed a genetic test for IRD prior to or at the date of inclusion. Patients who had been prescribed a genetic test for IRD prior to or at the date of inclusion. Patients who present at least one of the following non-inclusion criteria cannot be included in this study: Patients/Parents/Legally authorized representatives (LAR opposed to the collection and processing of their medical data/the medical data of their children/the medical data of the person for whom they are LAR; Patients/Parents/Legally authorized representatives (LAR refusing genetic testing): Patients who are suffering from any other retinal disorder on optic neuropathy that may clinically or genetically overlay with IRD or non-genetic (phenocopy); Patients/parents/Legally authorized representatives (LAR refusing genetic testing): Patients (paking decision-making capacity: Menta incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation. French reference and competence centers for rare eye diseases an gathered within the SENSGENE network. The Filière de sant maladies rares (FSMR) SENSGENE network. The Filière de sant maladies rares | | |
| with IRD or with high suspicion for IRDs based on clinica examination and functional tests (such as fundus exam an ERG), regardless of genetic testing Patients who attended a consultation at one of the participating centers from SENSGENE network over the inclusion period starting from sites initiation Patients who had been prescribed a genetic test for IRD priod to or at the date of inclusion. Patients who present at least one of the following non-inclusion criteria cannot be included in this study: Patients/Parents/Legally authorized representatives (LAR opposed to the collection and processing of their medical data of their children/the medical data (the person for whom they are LAR; Patients who are suffering from any other retinal disorder on optic neuropathy that may clinically or genetically overlay with IRD or non-genetic (phenocopy); Patients/parents/Legally authorized representatives (LAR refusing genetic testing; Patients lacking decision-making capacity: Menta incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation. French reference and competence centers for rare eye diseases an gathered within the SENSGENE fulfills national missions around rare sensory diseases with the aim of improving the care of patients coordinating and encouraging research and developing training and information. Seven French reference and competence centers for the SENSGENE network will be contacted to participate in the study Conduct of the study Five coordinating or constitutive reference enters for rare eye diseases: HU-Necker-Enfants Malades-APHP (Paris), CHNO XV-XX (Paris), CHI Créteil, HU Strasbourg, CHU Montpelier. This study will set up a registry that will include all eligible patient with IRD who attended a consultation at one of the participatin, with IRD who attended a consultation at one of the participatin, with IRD who attended a consultation at one of the participatin, with IRD who attended a consultation at one of the participatin, with IRD who attended a co | | Only the patients who meet <u>all</u> the following inclusion criteria can be included in this study: |
| Patients who attended a consultation at one of the participating centers from SENSGENE network over the inclusion period starting from sites initiation Patients who had been prescribed a genetic test for IRD prior to or at the date of inclusion. Patients who present at least one of the following non-inclusion criteria cannot be included in this study: Patients/Parents/Legally authorized representatives (LAR opposed to the collection and processing of their medical data/the medical data of their children/the medical data/the medical data of their children/the medical data of the person for whom they are LAR; Patients who are suffering from any other retinal disorder of optic neuropathy that may clinically or genetically overlay with IRD or non-genetic (phenocopy); Patients/parents/Legally authorized representatives (LAR refusing genetic testing); Patients lacking decision-making capacity: Mental incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation. French reference and competence centers for rare eye diseases and gathered within the SENSGENE fulfills national missions around rare sensory diseases with the aim of improving the care of patients coordinating and encouraging research and developing training and information. Seven French reference and competence centers from the SENSGENE network will be contacted to participate in the study Five coordinating or constitutive reference centers for rare eye diseases: HU-Necker-Enfants Malades-APHP (Paris), CHNO XV-XX (Paris), CHI Créteil, HU Strasbourg, CHU Montpelier. This study will set up a registry that will include all eligible patient with IRD who attended a consultation at one of the participatin, with IRD who attended a consultation at one of the participatin. | | All patients, whatever age or gender, clinically diagnosed with IRD or with high suspicion for IRDs based on clinical examination and functional tests (such as fundus exam and FRG), regardless of genetic testing. |
| Patients who had been prescribed a genetic test for IRD prio to or at the date of inclusion. Patients who present at least one of the following non-inclusion criteria cannot be included in this study: Patients/Parents/Legally authorized representatives (LAR opposed to the collection and processing of their medical data/the medical data of their children/the medical data of the children/the medical data of the person for whom they are LAR; Patients who are suffering from any other retinal disorder or optic neuropathy that may clinically or genetically overlay with IRD or non-genetic (phenocopy); Patients/parents/Legally authorized representatives (LAR refusing genetic testing; Patients lacking decision-making capacity: Menta incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation. French reference and competence centers for rare eye diseases and gathered within the SENSGENE network. The Fillère de sant maladies rares (FSMR) SENSGENE fulfills national missions around rare sensory diseases with the aim of improving the care of patients coordinating and encouraging research and developing training and information. Seven French reference and competence centers from the SENSGENE network will be contacted to participate in the study Conduct of the study Five coordinating or constitutive reference centers for rare eye diseases: HU-Necker-Enfants Malades-APHP (Paris), CHNO XV-XX (Paris), CHI Créteil, HU Strasbourg, CHU Montpelier. Time to competence centers for rare eye diseases: CHU Nantes and CHU Lille This study will set up a registry that will include all eligible patient with IRD who attended a consultation at one of the participation. | | <ul> <li>Patients who attended a consultation at one of the<br/>participating centers from SENSGENE network over the</li> </ul> |
| criteria cannot be included in this study: Patients/Parents/Legally authorized representatives (LAR opposed to the collection and processing of their medica data/the medical data of their children/the medical data of their children/the medical data of the person for whom they are LAR; Patients who are suffering from any other retinal disorder of optic neuropathy that may clinically or genetically overlay with IRD or non-genetic (phenocopy); Patients/parents/Legally authorized representatives (LAR refusing genetic testing; Patients lacking decision-making capacity: Menta incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation. French reference and competence centers for rare eye diseases an gathered within the SENSGENE network. The Filière de sant maladies rares (FSMR) SENSGENE fulfills national missions around rare sensory diseases with the aim of improving the care of patients coordinating and encouraging research and developing training and information. Seven French reference and competence centers from the SENSGENE network will be contacted to participate in the study Conduct of the study Five coordinating or constitutive reference centers for rare eye diseases: Hu-Necker-Enfants Malades-APHP (Paris), CHNO XV-XX (Paris), CHI Créteil, HU Strasbourg, CHU Montpelier. Two competence centers for rare eye diseases: CHU Nantes and CHU Lille This study will set up a registry that will include all eligible patient with IRD who attended a consultation at one of the participating with IRD who attended a consultation at one | | Patients who had been prescribed a genetic test for IRD prior |
| opposed to the collection and processing of their medical data/the medical data of their children/the medical data of the children/the medical data of the person for whom they are LAR; • Patients who are suffering from any other retinal disorder of optic neuropathy that may clinically or genetically overlay with IRD or non-genetic (phenocopy); • Patients/parents/Legally authorized representatives (LAR refusing genetic testing; • Patients lacking decision-making capacity: Menta incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation. French reference and competence centers for rare eye diseases are gathered within the SENSGENE fulfills national missions around rare sensory diseases with the aim of improving the care of patients coordinating and encouraging research and developing training and information. Seven French reference and competence centers from the SENSGENE network will be contacted to participate in the study • Five coordinating or constitutive reference centers for rare eye diseases: HU-Necker-Enfants Malades-APHP (Paris), CHNO XV-XX (Paris), CHI Créteil, HU Strasbourg, CHU Montpelier. • Two competence centers for rare eye diseases: CHU Nantes and CHU Lille This study will set up a registry that will include all eligible patient with IRD who attended a consultation at one of the participating at th | Inclusion and non-inclusion criteria | Patients who present <u>at least one</u> of the following non-inclusion criteria cannot be included in this study: |
| optic neuropathy that may clinically or genetically overlar with IRD or non-genetic (phenocopy); • Patients/parents/Legally authorized representatives (LAR refusing genetic testing; • Patients lacking decision-making capacity: Mental incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation. French reference and competence centers for rare eye diseases are gathered within the SENSGENE network. The Filière de sant maladies rares (FSMR) SENSGENE fulfills national missions around rare sensory diseases with the aim of improving the care of patients coordinating and encouraging research and developing training and information. Seven French reference and competence centers from the SENSGENE network will be contacted to participate in the study • Five coordinating or constitutive reference centers for rare eye diseases: HU-Necker-Enfants Malades-APHP (Paris), CHNO XV-XX (Paris), CHI Créteil, HU Strasbourg, CHU Montpelier. • Two competence centers for rare eye diseases: CHU Nantes and CHU Lille This study will set up a registry that will include all eligible patient with IRD who attended a consultation at one of the participating with IRD who att | | opposed to the collection and processing of their medical data/the medical data of their children/the medical data of the person for whom they are LAR; |
| Patients/parents/Legally authorized representatives (LAR refusing genetic testing; Patients lacking decision-making capacity: Menta incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation. French reference and competence centers for rare eye diseases are gathered within the SENSGENE network. The Filière de santimaladies rares (FSMR) SENSGENE fulfills national missions around rare sensory diseases with the aim of improving the care of patients coordinating and encouraging research and developing training and information. Seven French reference and competence centers from the SENSGENE network will be contacted to participate in the study Five coordinating or constitutive reference centers for rare eye diseases: HU-Necker-Enfants Malades-APHP (Paris), CHNO XV-XX (Paris), CHI Créteil, HU Strasbourg, CHU Montpelier. Two competence centers for rare eye diseases: CHU Nantes and CHU Lille This study will set up a registry that will include all eligible patient with IRD who attended a consultation at one of the participating with IRD who attended a consultation at one of the partici | | optic neuropathy that may clinically or genetically overlap |
| incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation. French reference and competence centers for rare eye diseases are gathered within the SENSGENE network. The Filière de sant maladies rares (FSMR) SENSGENE fulfills national missions around rare sensory diseases with the aim of improving the care of patients coordinating and encouraging research and developing training and information. Seven French reference and competence centers from the SENSGENE network will be contacted to participate in the study • Five coordinating or constitutive reference centers for rare eye diseases: HU-Necker-Enfants Malades-APHP (Paris), CHNO XV-XX (Paris), CHI Créteil, HU Strasbourg, CHU Montpelier. • Two competence centers for rare eye diseases: CHU Nantes and CHU Lille This study will set up a registry that will include all eligible patient with IRD who attended a consultation at one of the participating | | Patients/parents/Legally authorized representatives (LAR) |
| gathered within the SENSGENE network. The Filière de sante maladies rares (FSMR) SENSGENE fulfills national missions around rare sensory diseases with the aim of improving the care of patients coordinating and encouraging research and developing training and information. Seven French reference and competence centers from the SENSGENE network will be contacted to participate in the study • Five coordinating or constitutive reference centers for rare eye diseases: HU-Necker-Enfants Malades-APHP (Paris), CHNO XV-XX (Paris), CHI Créteil, HU Strasbourg, CHU Montpelier. • Two competence centers for rare eye diseases: CHU Nantes and CHU Lille This study will set up a registry that will include all eligible patient with IRD who attended a consultation at one of the participating | | incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation. |
| rare sensory diseases with the aim of improving the care of patients coordinating and encouraging research and developing training and information. Seven French reference and competence centers from the SENSGENE network will be contacted to participate in the study • Five coordinating or constitutive reference centers for rare eye diseases: HU-Necker-Enfants Malades-APHP (Paris), CHNO XV-XX (Paris), CHI Créteil, HU Strasbourg, CHU Montpelier. • Two competence centers for rare eye diseases: CHU Nantes and CHU Lille This study will set up a registry that will include all eligible patient with IRD who attended a consultation at one of the participating | | French reference and competence centers for rare eye diseases are gathered within the SENSGENE network. The Filière de santé |
| Five coordinating or constitutive reference centers for rare eye diseases: HU-Necker-Enfants Malades-APHP (Paris), CHNO XV-XX (Paris), CHI Créteil, HU Strasbourg, CHU Montpelier. Two competence centers for rare eye diseases: CHU Nantes and CHU Lille This study will set up a registry that will include all eligible patient with IRD who attended a consultation at one of the participating | Conduct of the study | maladies rares (FSMR) SENSGENE fulfills national missions around rare sensory diseases with the aim of improving the care of patients, coordinating and encouraging research and developing training and information. Seven French reference and competence centers from the SENSGENE network will be contacted to participate in the study. |
| Nantes and CHU Lille This study will set up a registry that will include all eligible patient with IRD who attended a consultation at one of the participating | | CHNO XV-XX (Paris), CHI Créteil, HU Strasbourg, CHU<br>Montpelier. |
| Required sample size with IRD who attended a consultation at one of the participating | | |
| | Required sample size | This study will set up a registry that will include all eligible patients with IRD who attended a consultation at one of the participating centers from SENSGENE network. |



For the Cross-sectional registry no sample size calculation is required as this registry will record patient fulfilling the sets of criteria defined and will allow to have an estimation of the target population at the national level.

Given the capacity of sites to screen patients over one year (around 3000 patients), the inclusion of patients into the study will be limited to the first 1000 patients in order to favor the data collection quality by limiting the sites workload. This will encourage the inclusion of the patients exhaustively, especially for high volume sites for which this registry represents a deep work. However, it should be reminded that this study is a starter study that is planned to be extended to a larger national registry.

The precision can be estimated for a sample size of 1000 patients while considering 5% loss (patients not evaluable for the primary objective or not meeting all selection criteria).

The following table presents the precision and the corresponding 2-sided 95% confidence interval (CI) to describe the distribution of IRD type (proportions varying from 10% to 50% for each modality) and a sample size of 1000 patients.

Table. Precision and corresponding 2-sided 95% CI given the proportion of a modality varying from 10% to 50% and a sample size of 1000 patients (5% of non-evaluable patients)

| | Proportion | | | | |
|---|---|---|---|---|---|
| | 10% | 20% | 30% | 40% | 50% |
| n | Precision | Precision | Precision | Precision | Precision |
| Précision<br>(%) | 1.9 | 2.5 | 2.9 | 3.1 | 3.2 |
| 95% CI | 8.1; 11.9 | 17.5; 22.5 | 27.1; 32.9 | 36.9; 43.1 | 46.8; 53.2 |

The precision (e) is calculated based on the normal approximation using the following formula:

$$e = \sqrt{\frac{1,96^2 * (p - p^2)}{n}}$$

where p is the proportion of a given modality and n is the number of patients.

## Statistical method

A descriptive analysis will be conducted on all study endpoints for which data has been collected both for the overall study population and per subgroups of interest where relevant (e.g. patients' clinical characteristics, classification (class 4 and 5), nature of the mutation, the values of visual acuity (VA) and visual field (VF), date of genetic testing, clinical phenotype, type of genetic analysis performed and unsolved patients) as long as that the sizes of the sub-groups are relevant for statistical estimations. The subgroups' modalities and associated endpoints will be detailed in the Statistical Analysis Plan.

The following statistics will be provided for quantitative variables: number and proportion of patients with non-missing and missing



| | values per variable, mean, standard deviation (StD), median, first quartile (Q1), third quartile (Q3), minimum and maximum value, the mode (especially for discrete quantitative variables with limited variability). |
|---|---|
| | For qualitative variables, the number and proportion of each variable modality will be provided together with the number of missing values. Proportion will be computed based on the population with non-missing data. |
| | Exploratory comparison between study subgroups might be considered. Statistical tests will be based on the type and distribution of the variables. All comparison tests will be two-tailed with a standard type 1 error threshold of 5% (significance level). |
| | The enrollment of patients in the study will be limited to a maximum of 1000 patients, registered over a variable period of time limited to 12 months. |
| | This study design therefore presents bias related to the heterogeneous duration of patients' inclusion which depends on the activity size of each participating physician. |
| | In order to take into account the biases associated with this study design and be able to extrapolate results at the national level, an adjustment is planned for descriptive analyses over the registry using a weight applied at center level. |
| Expected benefits | Implementation of an IRD national registry including all data related to IRD and presenting their clinical features may help to deepen the epidemiologic and genetics knowledge of IRDs. No direct benefit to the participating patient is expected from this study but the knowledge generated from this study may benefit future patients. |
| Drovisional schodule | -Maximum duration of the inclusion phase: 12 months or themaximum of 1000 patients is reached, whatever occurs first (a) -Maximum duration of participation of each patient: 12months (b) -Maximum total duration of the study: 24 months (= a+b) |
| Provisional schedule | -Exclusion from other interventional studies while patientsparticipate to the present clinical trial: None -End of trial: The study end corresponds to the end of the collection of gene testing results of the participation of the last subject in the study. |